CLINICAL TRIAL: NCT02143362
Title: Dexmedetomidine Combined With the Closed Loop of Target Controlled Infusion of Propofol for Anesthesia With Intraoperative Wake Up-single Center,Random,Controlled Trial
Brief Title: Dexmedetomidine Combined With the Closed Loop of Target Controlled Infusion of Propofol for Anesthesia With Intraoperative Wake up
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dex anesthesia
Record Dates: First submitted 2014-05-15; First posted 2014-05-21 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Anesthesia; Reaction
Keywords: Intraoperative wake up; Closed loop of target controlled infusion; Dexmedetomidine; Propofol
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine group (Experimental): 1. Infusion of dexmedetomidine(0.8μg/kg) at10 minutes before anesthesia induction.
  2. Infusion of dexmedetomidine at 0.4 μg•kg-1•h-1during anesthesia maintenance.
  3. The infusion rate of dexmedetomidine was reduced to 0.1 μg•kg-1•h-1 for awaken test.
  Interventions: Drug: Anesthesia induction,propofol, remifentanil ,cisatracurium; Drug: Anesthesia maintenance , propofol,remifentanil,cisatracurium; Procedure: Awaken test
- Control group (Placebo Comparator): 1. Infusion normal saline(0.8μg/kg) at 10 minutes before anesthesia induction.
  2. Infusion normal saline at 0.4 μg•kg-1•h-1 during anesthesia maintenance.
  3. The infusion rate of normal saline was reduced to 0.1 μg•kg-1•h-1 for awaken test.
  Interventions: Drug: Anesthesia induction,propofol, remifentanil ,cisatracurium; Drug: Anesthesia maintenance , propofol,remifentanil,cisatracurium; Procedure: Awaken test

INTERVENTIONS:
Drug: Anesthesia induction,propofol, remifentanil ,cisatracurium — 1. Target Controlled Infusion propofol and remifentanil to targeted plasma concentrations are 4 μg/ ml and 4 ng/ml respectively.
  2. Intermittent injection cisatracurium (0.15mg/kg).
  3. A laryngeal mask airway will be placed when bispectral electroencephalogram index is reduced to 60.
Drug: Anesthesia maintenance , propofol,remifentanil,cisatracurium — 1. Closed-loop target controlled infusion of propofol ,Bispectral electroencephalogram index feedback value will be set at 50.
  2. Target Controlled Infusion remifentanil , targeted plasma concentrations are 3~6ng/ml ,maintain heart rate to 60~100 beats per minute and mean blood pressure to 70~105 mmHg.
  3. Intermittent injection cisatracurium (0.05mg/kg).
Procedure: Awaken test — 1. Stopped Closed-loop target controlled infusion of cisatracurium and propofol 30 minutes before awaken test.
  2. In dexmedetomidine group,dexmedetomidine infusion rate will be reduced to 0.1 μg•kg-1•h-1. In control group ,normal saline infusion will be given with the same infusion rate as dexmedetomidine group .
  3. Call patients' name and require them to move both feet every 30 seconds after patients recovered normal respiration.
  4. Patients will be considered to be awake when recover normal respiration and make responsive to verbal commands correctly .
  5. Patients will receive initial anesthesia after finish awaken test.

SUMMARY:
The study designed to explore the efficacy and safety of the closed loop of target controlled infusion dexmedetomidine combined with propofol for anesthesia with intraoperative wake up.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Ongoing brain functional area surgery with intraoperative wake up.
* American Society of Anesthesiologists class I to II.
* Aged between 18 and 65 years old.
* Weight between plus or minus 20% of the standard weight. Male: (height cm - 80) × 70% = standard weight Female: (height cm - 70) × 60% = standard weight

Exclusion Criteria:

* History of hypertension.
* Serious heart,brain,liver,kidney, pulmonary, and endocrine disease or serious infection.
* Mental disability or mental disease.
* Use of sedative drug.
* Suspected or confirmed long term use of narcotic analgesics.
* Inability to exchange.
* Suspected or confirmed difficult airway.
* Suspected of malignant hyperthermia.
* Neuromuscular disease.
* Allergic to investigational products or with other contraindication.
* Subjects who are breastfeeding or pregnant.
* Participated in other study within 30 days .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of awaken test | The whole time of surgery,about 8 hours
The time from starting to awaken test to patient wakes up | From starting to awaken test to patient wakes up,about 3 hours
Blood sugar concentration | 30 minutes prior to awaken test,the moment of awake,5 minutes after awake,the moment after finish awaken test,10minutes after finish awaken test
Cortisol concentration | 30 minutes prior to awaken test,the moment of awake,5 minutes after awake,the moment after finish awaken test,10minutes after finish awaken test
Epinephrine concentration | 30 minutes prior to awaken test,the moment of awake,5 minutes after awake,the moment after finish awaken test,10minutes after finish awaken test
Norepinephrine concentration | 30 minutes prior to awaken test,the moment of awake,5 minutes after awake,the moment 30 minutes prior to awaken test,the moment of awake,5 minutes after awake,the moment after finish awaken test,10minutes after finish awaken test

SECONDARY OUTCOMES:
The duration of anesthesia from baseline to patient wake up | From baseline to patient wake up ,about 3 hours
The dosage of Cisatracurium before patient wakes up | From starting to awaken test to patient wakes up,about 3 hours
The dosage of propofol before patient wakes up | From starting to awaken test to patient wakes up,about 3 hours
The dosage of remifentanil before patient wakes up | From starting to awaken test to patient wakes up,about 3 hours
Heart rate | 30 minutes prior to awaken test,the moment of awake,5 minutes after awake,the moment after finish awaken test,10minutes after finish awaken test
Mean arterial pressure | 30 minutes prior to awaken test,the moment of awake,5 minutes after awake,the moment after finish awaken test,10minutes after finish awaken test
Bispectral electroencephalogram index | 30 minutes prior to awaken test,the moment of awake,5 minutes after awake,the moment after finish awaken test,10minutes after finish awaken test